CLINICAL TRIAL: NCT06843369
Title: Relation Between Inflammatory Responses and Sequelae of Pediatric Corrosive Ingestion Cases at Assiut University Hospitals
Brief Title: Relation Between Inflammatory Responses and Sequelae of Pediatric Corrosive Ingestion Cases in Assiut
Acronym: corrosive
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Mohamed Gamal Hassan, demonstrator ( Principal Investigator), Assiut University
Other Study IDs: corrosive ingestion cases
Record Dates: First submitted 2025-02-14; First posted 2025-02-25 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Corrosive Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: inflammatory markers — Serum amyloid A , cbc and IL-10

SUMMARY:
1. Evaluation of corrosive ingestion cases presented to Assiut university hospitals .
2. To assess the role of leukocytic parameters and inflammatory mediators in determining the severity of pediatric corrosive injuries and their correlation with long-term outcomes.

DETAILED DESCRIPTION:
Inflammatory response plays a vital role in the development of gastrointestinal complications following corrosive ingestion. Leucocytic parameters: neutrophil-to-lymphocyte ratio (NLR), neutrophils count and lymphocytic count from the peripheral blood, has emerged as an easily obtainable biomarker of acute inflammation .

Inflammatory mediators play a significant role in the body's response to injury. They also have a major impact on the pathophysiology of caustic injury, as they modulate the inflammatory response and tissue damage following exposure to corrosive substances. Therefore, they can potentially serve as prognostic biomarkers to assess the severity of caustic injury .

Acute phase reactants (APR) are inflammatory markers that exhibit significant changes in serum concentration during inflammation. These are also important mediators produced in the liver during acute and chronic inflammatory states. Their concentrations increase during inflammation. Serum amyloid A protein (SAA) is a pro-inflammatory mediator, and its concentration can increase from healthy levels of less than 3 mg per liter to more than 1000 mg per liter in the presence of inflammation, and it can remain elevated for as long as the inflammatory disease remains active .

Interleukin 10 (IL-10) is an anti-inflammatory cytokine that plays a crucial role in preventing inflammatory diseases, that generally begins to increase within a few hours after the onset of injury, although its peak may not occur until later (usually within 24-48 hours). Its release is often a part of the body's feedback mechanism to balance the acute inflammatory response .

DROOL caustic ingestion score is a diagnostic tool used to evaluate patients with corrosive ingestion through these parameters: drooling, dysphagia, oropharyngeal burns, others (fever, hematemesis, abdominal tenderness) and leukocytosis. It ranges from 0 to 10, with the best score being 10 .

ELIGIBILITY:
Inclusion Criteria:

* All cases diagnosed with corrosive ingestion presented at Assiut university hospital.

Exclusion Criteria:

* Cases with pre-existing inflammatory diseases
* Cases with emergencies other than corrosive ingestion.
* Patients with delay time more than 48hours.
* Pediatric cases whose legal guardians are unavailable or refuse to provide consent.

Max Age: 16 Years | Sex: All
Age Groups: Child
Study Population: Cases admitted to Assiut university hospitals with history of corrosive ingestion.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
correlation between inflammatory responses and sequelae of Pediatric Corrosive Ingestion cases at Assiut University Hospitals | march 2025 to February 2026
  Blood sample will be collected to measure Complete blood Count with differential leukocytic count in percent to assess the severity of inflammation in corrosive cases
assess the severity of corrosive ingestion cases clinically | march 2025 to February 2026
  through a questionnaire and DROOL corrosive ingestion score from 0 to 10 with 10 being the best score

CONTACTS AND LOCATIONS:
Overall Officials: hayam zakaria, prof dr, Study Director — Assiut University

REFERENCES:
- [Background] Cheng HT, Seak CJ, Cheng CC, Chen TH, Sung CM, Kang SC, Chen YJ, Ng CJ, Lee CW, Huang SW, Huang HC, Yen TH. Profiling of inflammatory cytokines in patients with caustic gastrointestinal tract injury. PLoS One. 2021 Nov 18;16(11):e0260012. doi: 10.1371/journal.pone.0260012. eCollection 2021. PMID 34793546
- [Background] Poonthottathil F, Suresh S, Nayer J, Aggarwal P. Diagnostic accuracy of drooling, reluctance, oropharynx, others, and leukocytosis score as a predictor of mortality and complications following acute corrosive ingestion. Turk J Emerg Med. 2023 Oct 3;23(4):225-231. doi: 10.4103/tjem.tjem_128_23. eCollection 2023 Oct-Dec. PMID 38024188